CLINICAL TRIAL: NCT02840851
Title: Brain Blood Flow Response to Hypercapnia in Healthy Adults: The Effect of Age and Sex
Brief Title: Brain Blood Flow: Age and Gender
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-0403; A176000 (Other: UW, Madison); EDUC/KINESIOLOGY/KINESIO (Other: UW, Madison)
Record Dates: First submitted 2016-07-19; First posted 2016-07-21 (Estimated); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Healthy; Aging
Keywords: Magnetic Resonance Imaging; Transcranial Doppler Ultrasound; Hypercapnia
MeSH Terms: conditions — Hypercapnia | interventions — Magnetic Resonance Imaging; Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Healthy young women: Healthy young women between the age of 20-34 years.
  Interventions: Device: MRI; Device: TCD
- Healthy young men: Healthy young men between the age of 20-34 years.
  Interventions: Device: MRI; Device: TCD
- Healthy older women: Healthy older women between the age of 50-64 years.
  Interventions: Device: MRI; Device: TCD
- Healthy older men: Healthy older men between the age of 50-64 years.
  Interventions: Device: MRI; Device: TCD

INTERVENTIONS:
Device: MRI — Participants will undergo a MRI scan while two stepwise CO2 elevations are applied to the participant by adding fractional concentration of inspired CO2 (FICO2) at 4% and 6% each time. The end tidal CO2 (PetCO2) will be elevated and maintained constant for a few minutes at each target level. Breath-by-breath changes in respiratory rate and PetCO2 will be measured.
  Other Names: Magnetic Resonance Imaging
Device: TCD — Participants will undergo a TCD scan while two stepwise CO2 elevations are applied to the participant by adding fractional concentration of inspired CO2 (FICO2) at 4% and 6% each time. The end tidal CO2 (PetCO2) will be elevated and maintained constant for a few minutes at each target level. Breath-by-breath changes in respiratory and PetCO2 will be measured.
  Other Names: Transcranial Doppler Ultrasound

SUMMARY:
Baseline cerebral blood flow through the middle cerebral artery (MCA) and cerebral vasodilator response of the MCA to inhaled carbon dioxide (CO2) will be measured in young women, young men, older women, and older men using Magnetic Resonance (MR) imaging and transcranial Doppler ultrasound (TCD). Data collection techniques will be compared.

DETAILED DESCRIPTION:
The investigators have recently shown that cerebral blood flow responses to chemical stimuli are reduced in healthy older adults. The investigators also have preliminary data suggesting that sex differences in cerebrovascular regulation exist. The overall goal of this application is to extend on the investigators previous studies by employing advanced neuroimaging techniques to enhance the investigators understanding of neurovascular coupling in healthy aging. This study will collect clinically significant data with implications for the future risk of cognitive decline and Alzheimer's disease.

The research aims are:

1. To determine the effect of age and sex on baseline cerebral blood flow through the middle cerebral artery (MCA).
2. To determine the effect of age and sex on cerebral vasodilator responses.
3. To determine if the cerebrovascular responses measured by transcranial Doppler ultrasound (TCD) are associated with the cerebrovascular responses measured by Magnetic Resonance (MR) imaging.

ELIGIBILITY:
Inclusion Criteria:

* Between 20-34 or 50-69 years
* Body mass index <34 kg/m2

Exclusion Criteria:

* Current smoker
* History or evidence of: hepatic disease, renal disease, hematological disease, peripheral vascular disease, stroke/neurovascular disease, diabetes, hypertension
* Part of a vulnerable population (e.g. pregnant women, prisoner, individuals lacking capacity to consent, etc.)
* Older females only: subject is not post-menopausal

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects for this study will include healthy young adults (20-34 years old) and healthy older adults (50-69 years old). Both men and women will be eligible to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Middle Cerebral Artery Blood Flow Measurement | 75 minutes
  Utilize the TCD and MR imaging to measure middle cerebral artery blood flow in the brain while the participant is at rest.
Middle Cerebral Artery Blood Flow Reactivity to Hypercapnia | 75 minutes
  Utilize the TCD and MR imaging to measure middle cerebral artery blood flow reactivity to hypercapnic gas.

CONTACTS AND LOCATIONS:
Overall Officials: Jill N Barnes, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Girouard H, Iadecola C. Neurovascular coupling in the normal brain and in hypertension, stroke, and Alzheimer disease. J Appl Physiol (1985). 2006 Jan;100(1):328-35. doi: 10.1152/japplphysiol.00966.2005. PMID 16357086
- [Background] Bakker SL, de Leeuw FE, den Heijer T, Koudstaal PJ, Hofman A, Breteler MM. Cerebral haemodynamics in the elderly: the rotterdam study. Neuroepidemiology. 2004 Jul-Aug;23(4):178-84. doi: 10.1159/000078503. PMID 15272220
- [Background] Selim M, Jones R, Novak P, Zhao P, Novak V. The effects of body mass index on cerebral blood flow velocity. Clin Auton Res. 2008 Dec;18(6):331-8. doi: 10.1007/s10286-008-0490-z. Epub 2008 Aug 22. PMID 18726054
- [Background] Dandona P, James IM, Newbury PA, Woollard ML, Beckett AG. Cerebral blood flow in diabetes mellitus: evidence of abnormal cerebrovascular reactivity. Br Med J. 1978 Jul 29;2(6133):325-6. doi: 10.1136/bmj.2.6133.325. PMID 687900
- [Background] Barnes JN, Schmidt JE, Nicholson WT, Joyner MJ. Cyclooxygenase inhibition abolishes age-related differences in cerebral vasodilator responses to hypercapnia. J Appl Physiol (1985). 2012 Jun;112(11):1884-90. doi: 10.1152/japplphysiol.01270.2011. Epub 2012 Mar 22. PMID 22442028
- [Background] Lipsitz LA, Mukai S, Hamner J, Gagnon M, Babikian V. Dynamic regulation of middle cerebral artery blood flow velocity in aging and hypertension. Stroke. 2000 Aug;31(8):1897-903. doi: 10.1161/01.str.31.8.1897. PMID 10926954
- [Background] Kearney-Schwartz A, Rossignol P, Bracard S, Felblinger J, Fay R, Boivin JM, Lecompte T, Lacolley P, Benetos A, Zannad F. Vascular structure and function is correlated to cognitive performance and white matter hyperintensities in older hypertensive patients with subjective memory complaints. Stroke. 2009 Apr;40(4):1229-36. doi: 10.1161/STROKEAHA.108.532853. Epub 2009 Feb 26. PMID 19246701
- [Background] Smith EE, Greenberg SM. Beta-amyloid, blood vessels, and brain function. Stroke. 2009 Jul;40(7):2601-6. doi: 10.1161/STROKEAHA.108.536839. Epub 2009 May 14. PMID 19443808
- [Background] Celermajer DS, Sorensen KE, Bull C, Robinson J, Deanfield JE. Endothelium-dependent dilation in the systemic arteries of asymptomatic subjects relates to coronary risk factors and their interaction. J Am Coll Cardiol. 1994 Nov 15;24(6):1468-74. doi: 10.1016/0735-1097(94)90141-4. PMID 7930277
- [Background] Panza JA, Quyyumi AA, Brush JE Jr, Epstein SE. Abnormal endothelium-dependent vascular relaxation in patients with essential hypertension. N Engl J Med. 1990 Jul 5;323(1):22-7. doi: 10.1056/NEJM199007053230105. PMID 2355955
- [Background] Kugiyama K, Kerns SA, Morrisett JD, Roberts R, Henry PD. Impairment of endothelium-dependent arterial relaxation by lysolecithin in modified low-density lipoproteins. Nature. 1990 Mar 8;344(6262):160-2. doi: 10.1038/344160a0. PMID 2106627
- [Background] Luscher TF, Diederich D, Siebenmann R, Lehmann K, Stulz P, von Segesser L, Yang ZH, Turina M, Gradel E, Weber E, et al. Difference between endothelium-dependent relaxation in arterial and in venous coronary bypass grafts. N Engl J Med. 1988 Aug 25;319(8):462-7. doi: 10.1056/NEJM198808253190802. PMID 3136329
- [Background] Mitchell GF, van Buchem MA, Sigurdsson S, Gotal JD, Jonsdottir MK, Kjartansson O, Garcia M, Aspelund T, Harris TB, Gudnason V, Launer LJ. Arterial stiffness, pressure and flow pulsatility and brain structure and function: the Age, Gene/Environment Susceptibility--Reykjavik study. Brain. 2011 Nov;134(Pt 11):3398-407. doi: 10.1093/brain/awr253. PMID 22075523
- [Background] Ide K, Eliasziw M, Poulin MJ. Relationship between middle cerebral artery blood velocity and end-tidal PCO2 in the hypocapnic-hypercapnic range in humans. J Appl Physiol (1985). 2003 Jul;95(1):129-37. doi: 10.1152/japplphysiol.01186.2002. PMID 19278048
- [Background] Ivancev V, Bakovic D, Obad A, Breskovic T, Palada I, Joyner MJ, Dujic Z. Effects of indomethacin on cerebrovascular response to hypercapnea and hypocapnea in breath-hold diving and obstructive sleep apnea. Respir Physiol Neurobiol. 2009 May 15;166(3):152-8. doi: 10.1016/j.resp.2009.03.001. Epub 2009 Mar 18. PMID 19442931
- [Background] Xie A, Skatrud JB, Morgan B, Chenuel B, Khayat R, Reichmuth K, Lin J, Dempsey JA. Influence of cerebrovascular function on the hypercapnic ventilatory response in healthy humans. J Physiol. 2006 Nov 15;577(Pt 1):319-29. doi: 10.1113/jphysiol.2006.110627. Epub 2006 Aug 24. PMID 16931556
- [Background] Mendelsohn ME, Karas RH. The protective effects of estrogen on the cardiovascular system. N Engl J Med. 1999 Jun 10;340(23):1801-11. doi: 10.1056/NEJM199906103402306. No abstract available. PMID 10362825
- [Background] Newell DW, Aaslid R, Lam A, Mayberg TS, Winn HR. Comparison of flow and velocity during dynamic autoregulation testing in humans. Stroke. 1994 Apr;25(4):793-7. doi: 10.1161/01.str.25.4.793. PMID 7909175
- [Background] Coverdale NS, Badrov MB, Shoemaker JK. Impact of age on cerebrovascular dilation versus reactivity to hypercapnia. J Cereb Blood Flow Metab. 2017 Jan;37(1):344-355. doi: 10.1177/0271678X15626156. Epub 2016 Jan 12. PMID 26759432
- [Derived] Miller KB, Howery AJ, Rivera-Rivera LA, Johnson SC, Rowley HA, Wieben O, Barnes JN. Age-Related Reductions in Cerebrovascular Reactivity Using 4D Flow MRI. Front Aging Neurosci. 2019 Oct 17;11:281. doi: 10.3389/fnagi.2019.00281. eCollection 2019. PMID 31680935